CLINICAL TRIAL: NCT03269539
Title: Assessment of Siemens' GoBrain and DotBrain Software
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: University of Saskatchewan (Other)
Responsible Party: Sponsor
Other Study IDs: Bio 16-278
Record Dates: First submitted 2017-08-29; First posted 2017-08-31 (Actual); Last update posted 2017-08-31 (Actual); Status verified 2017-08

CONDITIONS: Headache
MeSH Terms: conditions — Headache

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Headache Patients: Patients Referred for MRI with History of Headaches
  Interventions: Other: MRI Imaging
- Motion prone patients: Patients without the ability to remain still for the entire protocol
  Interventions: Other: MRI Imaging

INTERVENTIONS:
Other: MRI Imaging

SUMMARY:
Our main approach in this research is to collect MR data using both a "Routine" and "Fast" brain protocol on the 3 Tesla Siemens Skyra scanner using a 20-Channel Head/Neck Coil to determine if the "Fast" protocol can collect data in less time without compromising patient care.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred for MRI with History of Headaches

Exclusion Criteria:

* Patient does not meet MRI safety criteria
* Patient has known Brain Pathology

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients referred for MRI with History of Headaches
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2016-11; Primary Completion 2017-11 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
Assessment of Siemens' GoBrain and DotBrain Software | 1 year

IPD SHARING:
Plan to Share IPD: No